CLINICAL TRIAL: NCT02272803
Title: A Phase 2, Randomized, Open Label Trial of Lenalidomide/Dexamethasone With or Without Elotuzumab in Subjects With Previously Untreated Multiple Myeloma in Japan
Brief Title: Phase II Study of Lenalidomide/Dexamethasone With or Without Elotuzumab for Newly Diagnosed MM Patients in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-116
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) (Experimental): Drug: Lenalidomide
  Capsules, Oral, 25 mg, once daily, on Days 1-21, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Drug: Dexamethasone
  Tablets, Oral 28 mg and Intravenous (IV) 8 mg, once daily, on Days 1, 8, 15, 22 (cycles 1&2) ; Days 1 &15 (cycles 3-18); Day 1 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Tablets, Oral, 40 mg, once daily, on Days 8 & 22 (cycles 3-18); Days 8, 15, 22 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Biological: Elotuzumab (BMS-901608)
  Solution, Intravenous (IV), 10 mg/kg, weekly, on Days 1, 8, 15, 22 (cycles 1&2); Days 1 and 15 (cycles 3-18), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Solution, Intravenous (IV), 20 mg/kg, Day 1 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Biological: Elotuzumab (BMS-901608)
- Arm B: Lenalidomide + Dexamethasone (Active Comparator): Drug: Lenalidomide
  Capsules, Oral, 25 mg, once daily, on Days 1-21, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Drug: Dexamethasone
  Tablets, Oral, 40 mg, weekly, on Days 1, 8, 15, 22, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide
Drug: Dexamethasone
Biological: Elotuzumab (BMS-901608)
  Arms: Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608)

SUMMARY:
The purpose of this study is to determine the efficacy of Lenalidomide/Dexamethasone + Elotuzumab in the subjects with newly diagnosed, previously untreated Multiple Myeloma (MM) in Japan.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Newly diagnosed with symptomatic Multiple Myeloma (MM)
* Have not received any prior systemic anti-myeloma therapy
* Have measurable disease
* Are not candidates for high-dose therapy plus stem-cell transplantation (SCT) because of age (≥ 65 years) or coexisting conditions. Refusal to undergo high dose therapy with SCT is NOT sufficient for entry onto CA204-116 for a subject < 65 years old. There must be a comorbidity that prevents SCT for a subject < 65 years old

Exclusion Criteria:

* Non-secretory myeloma
* Smoldering MM, defined as asymptomatic MM with absence of lytic bone lesions
* Monoclonal Gammopathy of Undetermined Significance (MGUS)
* Active plasma cell leukemia
* Known Human Immunodeficiency Virus (HIV) infection or active hepatitis A, B, or C

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- Japan (26):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Aomori, Aomori
  - Local Institution, Chiba, Chiba
  - Local Institution, Kamogawa-shi, Chiba
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Maebashi, Gunma
  - Local Institution, Shibukawa-shi, Gunma
  - Local Institution, Fukuyama-shi, Hiroshima
  - Local Institution, Morioka, Iwate
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Niigata, Niigata
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Kawagoe-shi, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Utsunomiya, Tochigi
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Koto-ku, Tokyo
  - Local Institution, Shibuya-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Shinjuku-ku, Tokyo
  - Local Institution, Tachikawa-shi, Tokyo
  - Local Institution, Kasama-shi

REFERENCES:
- [Derived] Suzuki A, Kakugawa S, Miyoshi M, Hori M, Suzuki K, Furukawa Y, Ohta K. Soluble SLAMF7 is a predictive biomarker for elotuzumab therapy. Leukemia. 2020 Nov;34(11):3088-3090. doi: 10.1038/s41375-020-0860-7. Epub 2020 May 12. No abstract available. PMID 32398792
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 82 participants were randomized and treated.
Groups:
- Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608): Lenalidomide
  25 mg taken orally once daily, Days 1 - 21 of each cycle
  Dexamethasone
  Administered on Days 1, 8, 15, and 22 of each cycle:
  On weeks when elotuzumab is administered:
  * 28 mg taken orally (3 - 24 hours prior to start of elotuzumab infusion) AND
  * 8 mg IV (at least 45 minutes prior to elotuzumab administration)
  On weeks when elotuzumab is NOT administered:
  - 40 mg taken orally
  Elotuzumab (BMS-901608)
  * Cycle 1 - 2: 10 mg/kg IV, Days 1, 8, 15, 22
  * Cycle 3 - 18: 10 mg/kg IV, Days 1 and 15
  * Cycle 19 and beyond: 20 mg/kg IV, Day 1
- Arm B: Lenalidomide + Dexamethasone: Lenalidomide
  25 mg taken orally once a day, Days 1 - 21 of each cycle
  Dexamethasone
  40 mg taken orally, Days 1, 8, 15, and 22 of each cycle
Period: Overall Study
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) | Arm B: Lenalidomide + Dexamethasone
Started | 40 | 42
Completed | 0 | 0
Not Completed | 40 | 42
Not completed — Disease progression | 16 | 8
Not completed — Adverse Event unrelated to study drug | 3 | 5
Not completed — Study drug toxicity | 4 | 9
Not completed — Participant request to discontinue study treatment | 3 | 7
Not completed — Maximum clinical benefit | 4 | 2
Not completed — Poor/non-compliance | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 0 | 1
Not completed — Other reasons | 1 | 3
Not completed — Administrative reason by sponsor | 5 | 4

BASELINE CHARACTERISTICS:
Population: All treated particpants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) | Arm B: Lenalidomide + Dexamethasone | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All treated participants
  years | 72.6 (4.91) | 74.0 (6.32) | 73.3 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 23 | 20 | 43
    Male | 17 | 22 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 40 | 42 | 82
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Participants Treated With Elotuzumab + Lenalidomide/Dexamethasone (E-Ld)
Description: ORR is the proportion of randomized participants who achieve a stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or PR as determined by investigator using the International Myeloma Working Group (IMWG) response criteria.
  SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From first dose until documented response (assessed up to February 2017, approximately 24 months)
Population: Participants treated with E-Ld
Measure: Number (70% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608)
Number analyzed (Participants) | 40
Percentage of participants | 87.5 [79.7 to 92.9]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is the percentage of randomized participants who achieve a stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) as determined by investigator using the International Myeloma Working Group (IMWG) response criteria.
  SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From first dose until documented response, up to approximately 72 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) | Arm B: Lenalidomide + Dexamethasone
Number analyzed (Participants) | 40 | 42
Percentage of participants | 92.5 [79.6 to 98.4] | 73.8 [58.0 to 86.1]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of the first documented tumor progression, as determined by the investigator using the International Myeloma Working Group (IMWG) response criteria, or to death due to any cause, provided death does not occur more than 10 weeks (2 or more assessment visits) after the last tumor assessment. Clinical deterioration will not be considered progression.
Time Frame: From randomization to the date of first documented tumor progression or death due to any cause, up to approximately 72 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) | Arm B: Lenalidomide + Dexamethasone
Number analyzed (Participants) | 40 | 42
Months | NA [23.10 to NA] — Median and upper limit were not estimable due to an insufficient number of participants with events. | 43.33 [16.66 to NA] — Upper limit was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) vs Arm B: Lenalidomide + Dexamethasone; Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.41 to 1.67] — Hazard Ratio of E-Ld to Ld. Stratified by stage of disease (International Staging System 1 - 2 vs 3)

4. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: PFS rate is defined as the percentage of participants who have neither progressed nor died at the specified timepoints
Time Frame: From randomization up to the specified timepoints, up to 3 years
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) | Arm B: Lenalidomide + Dexamethasone
Number analyzed (Participants) | 40 | 42
Percentage of Participants
  1 year | 0.87 [0.72 to 0.95] | 0.89 [0.73 to 0.96]
  2 years | 0.67 [0.49 to 0.80] | 0.60 [0.41 to 0.75]
  3 years | 0.61 [0.42 to 0.75] | 0.56 [0.36 to 0.71]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 77 months). Serious Adverse events and other adverse events were assessed from date of first dose to 60 days following date of last dose (up to approximately 74 months).
Description: All randomized participants
Arm/Group | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) | Arm B: Lenalidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 2/40 | 6/42
Serious Adverse Events (participants affected / at risk) | 26/40 | 27/42
Other Adverse Events (participants affected / at risk) | 39/40 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) (N=40) | Arm B: Lenalidomide + Dexamethasone (N=42)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Eosinophilic myocarditis (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 7 | 7
Cataract subcapsular (Eye disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Ischaemic enteritis (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Disseminated varicella zoster virus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peri-implantitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 7
Pneumonia cryptococcal (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 1
C-reactive protein increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Lenalidomide + Dexamethasone + Elotuzumab (BMS-901608) (N=40) | Arm B: Lenalidomide + Dexamethasone (N=42)
Anaemia (Blood and lymphatic system disorders) | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 9 | 4
Lymphopenia (Blood and lymphatic system disorders) | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 11 | 9
Atrial fibrillation (Cardiac disorders) | 3 | 3
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2
Cataract (Eye disorders) | 17 | 12
Dry eye (Eye disorders) | 3 | 1
Glaucoma (Eye disorders) | 5 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Chronic gastritis (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 17 | 13
Dental caries (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 17 | 12
Haemorrhoids (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 6 | 5
Periodontal disease (Gastrointestinal disorders) | 1 | 3
Stomatitis (Gastrointestinal disorders) | 6 | 3
Vomiting (Gastrointestinal disorders) | 9 | 3
Malaise (General disorders) | 10 | 2
Non-cardiac chest pain (General disorders) | 3 | 1
Oedema (General disorders) | 2 | 3
Oedema peripheral (General disorders) | 12 | 12
Pyrexia (General disorders) | 17 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 8 | 1
Bronchitis (Infections and infestations) | 8 | 3
Cellulitis (Infections and infestations) | 2 | 3
Conjunctivitis (Infections and infestations) | 5 | 0
Cystitis (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 5 | 0
Gingivitis (Infections and infestations) | 2 | 3
Hepatitis B reactivation (Infections and infestations) | 3 | 0
Herpes virus infection (Infections and infestations) | 3 | 1
Herpes zoster (Infections and infestations) | 4 | 4
Influenza (Infections and infestations) | 5 | 2
Nasopharyngitis (Infections and infestations) | 18 | 18
Oral herpes (Infections and infestations) | 0 | 4
Osteomyelitis (Infections and infestations) | 1 | 3
Periodontitis (Infections and infestations) | 4 | 1
Pharyngitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 6 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Urinary tract infection (Infections and infestations) | 6 | 2
Contusion (Injury, poisoning and procedural complications) | 9 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 3
Blood creatinine increased (Investigations) | 2 | 4
C-reactive protein increased (Investigations) | 4 | 2
Creatinine renal clearance decreased (Investigations) | 6 | 0
Lymphocyte count decreased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 5 | 4
Platelet count decreased (Investigations) | 5 | 1
Weight decreased (Investigations) | 4 | 2
White blood cell count decreased (Investigations) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3
Dizziness (Nervous system disorders) | 4 | 6
Dysgeusia (Nervous system disorders) | 8 | 9
Headache (Nervous system disorders) | 6 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 3
Delirium (Psychiatric disorders) | 6 | 2
Insomnia (Psychiatric disorders) | 10 | 11
Chronic kidney disease (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 6
Purpura (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 12 | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT02272803/Prot_003.pdf
  • Statistical Analysis Plan (2017-04-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02272803/SAP_002.pdf